CLINICAL TRIAL: NCT05802017
Title: Relation Between Adverse Reactions to Food, Physical Performance and Health in a Mediterranean Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Marcela Gonzalez Gross, Prof. Dr., Universidad Politecnica de Madrid
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P2011600273
Record Dates: First submitted 2022-12-05; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Food Allergy; Food Intolerance; Adverse Reaction to Food
MeSH Terms: conditions — Food Hypersensitivity; Food Intolerance

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allergen-specific substitute diet (Experimental): Participants follow a 4-month allergen-specific diet according to their immunology results.
  Interventions: Other: Allergen-specific substitute diet
- Healthy diet (No Intervention): Participants follow a 4-month standard healthy diet.

INTERVENTIONS:
Other: Allergen-specific substitute diet — Substitution of IgG4 allergen-specific reactive foodstuffs for equivalent foodstuffs with similar nutritional value.
  Other Names: Substitute diet; IgG4 substitute diet
  Arms: Allergen-specific substitute diet

SUMMARY:
Since the prevalence of adverse reactions to foodstuffs (ARFS) has been steadily increasing and has become an alarming health concern, the general objective of this study is to analyze the prevalence of ARFS in Spanish adults of different physical condition.

DETAILED DESCRIPTION:
Individuals with associated diseases and symptomatology to ARFS will be selected and will be clinically and physically measured.

ELIGIBILITY:
Inclusion Criteria:

* Diseases and symptomatology associated to ARF.

Exclusion Criteria:

* Participation in other study.
* Pregnancy.
* Antibiotic treatment.
* Active Helicobacter pylori infection.
* Antidepressant, sleeping pill, or anxiolytic treatment.
* Job or lifestyle that potentially interferes with your regular sleep schedule.
* Active Cancer treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Immunoglobulin G4 and E response in subjects with subjective symptoms of adverse reactions to food. | 4-month intervention
  Immunoglobulin G4 and E reported in kilounits per liter through HELIA® Helmed Line Immunoassay.

SECONDARY OUTCOMES:
Body composition in sedentary and physically active population. | 4-month intervention
  Weight and Height will be combined to report BMI in kg/m^2 through Tanita equipment model MC-780MA.
Physical condition in sedentary and physically active population. | 4-month intervention
  Maximum rate of oxygen reported in VO₂max using GE Olmeda TuffSat®.
General health in subjects with subjective symptoms of adverse reactions to food. | 4-month intervention
  Health measured using number of cells reported in x10^6/mm^3 through spectrometry-flow cytometry Smty®.

CONTACTS AND LOCATIONS:
Overall Officials: Lisset S Pantoja Arevalo, MSc, Study Chair — Universidad Politecnica de Madrid; Marcela Gonzalez Gross, Prof Dr, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Facultad de Ciencias de la Actividad Física y del Deporte, Madrid, Spain

REFERENCES:
- [Derived] Pantoja-Arevalo L, Gesteiro E, Perez-Ruiz M, Lopez-Seoane J, Wusterhausen P, Matthias T, Urrialde R, Gonzalez-Gross M. The multifactorial approach and the food allergen-specific substitutive diet as a tool to manage and ameliorate adverse reactions to foodstuffs in adulthood: study protocol for a randomized controlled trial-the ALASKA study. Trials. 2024 Jul 20;25(1):494. doi: 10.1186/s13063-024-08307-2. PMID 39033266